CLINICAL TRIAL: NCT04506008
Title: Prospective Observational Trial of Two Neoadjuvant Hypofractionated Radiotherapy Regimens Followed by Surgical Resection in the Treatment of Soft Tissue Sarcomas
Brief Title: Hypofractionated Radiotherapy Followed by Surgical Resection in the Treatment of Soft Tissue Sarcomas
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Responsible Party: Principal Investigator, Eric Shinohara, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC SAR 2062
Record Dates: First submitted 2020-08-05; First posted 2020-08-10 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Soft Tissue Sarcomas
Keywords: Hypofractionated Radiotherapy
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group I (UH HRT) (Experimental): Patients undergo HRT daily for a total of 5 fractions followed by surgery.
  Interventions: Radiation: Ultra-Hypo-fractionation Radiotherapy; Procedure: Resection; Other: Questionnaire Administration
- Group II (MH HRT) (Experimental): Patients undergo HRT daily for a total of 15 fractions followed by surgery.
  Interventions: Procedure: Resection; Other: Questionnaire Administration; Radiation: Moderately-Hypo-fractionation Radiotherapy

INTERVENTIONS:
Radiation: Ultra-Hypo-fractionation Radiotherapy — Five fractions of pre-operative radiation
  Arms: Group I (UH HRT)
Procedure: Resection — Surgery
Other: Questionnaire Administration — Ancillary studies
Radiation: Moderately-Hypo-fractionation Radiotherapy — 15 fractions of pre-operative radiation
  Arms: Group II (MH HRT)

SUMMARY:
The trial will use neoadjuvant hypofractionated radiotherapy followed by surgical resection in the treatment for soft tissue sarcoma. It will allow patients to be treated over a shorter course (5 or 15 days of radiation) compared to the traditional 5 week regimen. It is proposed that this will be possible without increasing the risk of wound complication or local recurrence compared with a traditional 5 week course of pre-operative radiation.

DETAILED DESCRIPTION:
Study Objectives:

Primary:

* To investigate the efficacy of neoadjuvant hypo-fractionated radiotherapy (HRT) followed by surgical resection in the treatment of soft tissue sarcoma (STS) as measured by local control
* Examine the side effect profile using Radiation Therapy Oncology Group (RTOG) and Common Terminology Criteria for Adverse Events (CTCAE) acute and late side effects criteria and major and minor post-operative complication rates.

OUTLINE: Patients are assigned to 1 of 2 groups by the radiation oncologist.

GROUP I (ULTRA-HYPOFRACTIONATION [UH]): Patients undergo HRT daily for a total of 5 fractions followed by surgery.

GROUP II (MODERATE HYPOFRACTIONATION [MH]): Patients undergo HRT daily for a total of 15 fractions followed by surgery.

After completion of study treatment, patients are followed up within 3 months, then every 3-6 months for a minimum of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of a soft tissue sarcoma of extremity, pelvis, chest wall or trunk/abdominal wall (non-retroperitoneal location)
* ECOG performance status 0-2
* Patient must be deemed able to comply with radiation treatment and surgery

Exclusion Criteria:

* History of prior radiation to the same area to be irradiated
* Pregnancy
* Active collagen vascular disease or patients genetically predisposed to increased radiation related side effects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-02 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Local control rate | Approximately 2 years
  Will be estimated with a Beta-Binomial model with Beta(0.5, 0.5) as the prior distribution. The median and a 95% credible interval of the posterior distribution will be reported.

SECONDARY OUTCOMES:
Complication rate | Approximately 2 years
  The complication rate will be modeled with a Beta-Binomial model with Beta(0.5, 0.5) as the prior distribution, and it will be monitored continuously throughout the study. The complication rate will also be modeled with a Beta-Binomial model with Beta(0.5, 0.5) as the prior distribution, and it will be monitored continuously throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Shinohara, MD, Principal Investigator — Vanderbilt Medical Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/08/NCT04506008/ICF_000.pdf